CLINICAL TRIAL: NCT04176458
Title: Non-invasive Assessment of Liver Function in Patients Undergoing Heart and Liver Transplant Evaluation
Brief Title: Methacetin Breath Test in Patients With Liver Disease Secondary to Heart Disease
Acronym: MBT+Fontan
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: due to COVID 19 restrictions at our site
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Daniel Ganger, Principal Investigator, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STU00208318
Record Dates: First submitted 2019-02-12; First posted 2019-11-25 (Actual); Results first posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Dilated Cardiomyopathy; Tricuspid Atresia
MeSH Terms: conditions — Cardiomyopathy, Dilated; Tricuspid Atresia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- MBT in liver disease (Other): Methacetin Breath test (MBT) intervention. We will use the MBT test to measure time from administration of 13C methacetin to obtaining the peak elimination of 13CO2.
  Interventions: Device: Methacetin Breath Test (MBT)

INTERVENTIONS:
Device: Methacetin Breath Test (MBT) — The hypothesis is that MBT CPDR 20 in the Fontan patient is abnormal as a result of alterations in liver perfusion, liver cell metabolic capability and transhepatic resistance secondary to hemodynamics unique to the Fontan as well as end-organ liver damage. Due to lack of robust biomarkers or other risk stratification schemes, we aim to determine whether there is prognostic value in hepatic MBT CPDR 20 in the Fontan patient.

SUMMARY:
The aim of this project is assess a non-invasive functional liver tests in patients with the Fontan circulation that may be used for prognostic purposes. Specifically, we aim to determine whether there are alterations in Methacetin Breath Test (MBT) in the Fontan patient and if so, whether it is related to conventional tests of liver and cardiac function. The hypothesis is that MBT CPDR 20 in the Fontan patient is abnormal as a result of alterations in liver perfusion, liver cell metabolic capability and transhepatic resistance secondary to hemodynamics unique to the Fontan as well as end-organ liver damage. Due to lack of robust biomarkers or other risk stratification schemes, we aim to determine whether there is prognostic value in hepatic MBT CPDR 20 in the Fontan patient.

Aims - The aims of this study are three-fold:

1. To measure MBT parameter in a cohort of patients with Congestive (Dilated) Cardiomyopathy and a group of Fontan patients and compare results to published normal controls.
2. To explore any association between MBT parameter and clinical parameters already available, including Fontan hemodynamics as assessed by either of the following tests: cardiac catheterization, echocardiography, non-invasive imaging of the liver (CT or MRI), non-invasive assessment of liver stiffness (ARFI, MRE or Fibroscan), laboratory investigations, and clinical characteristics (i.e. age of patient, time since Fontan operation, type of Fontan etc.) within 12 months of the study.
3. To determine whether MBT is predictive of clinical outcomes: heart failure, clinically significant ascites, and time to transplant or death.

DETAILED DESCRIPTION:
Research Design and Methods Study Design: This is a prospective pilot cohort study in 20 patients with Dilated Congestive Cardiomyopathy (10) and a group of adult Fontan (10) recruited from an adult congenital heart disease clinic in a tertiary care center. Patients enrolled in the study will be prospectively followed for 3-5 years.

Study Timelines: We anticipate that it will take approximately 2 years to recruit patients who are to be included in this study. Patient will followed 3-5 years. However due to covid 19 issues recruitment did not go as planned and due to this delay we had to end study early. Since study terminated early, subjects will not be followed 3-5 years.

Study Endpoints: The aim of this project is assess a non-invasive functional liver tests in patients with the Fontan circulation that may be used for prognostic purposes.

PROCEDURES INVOLVED:

Methods Screening and consent Eligible patients will be screened and recruited through the outpatient Hepatology Clinic, Heart Failure Clinic and the Adult congenital heart disease clinic. They will be approached the day of the scheduled outpatient appointment by the PI or a study coordinator in a private room.

Informed consent will be obtained by the principal investigator, a sub-investigator or a member of the study team who is authorized to give consent. This will allow the potential subject sufficient opportunity to consider whether or not to participate and this will minimize the risk of influence or coercion. The subject will be informed of what the research entails. Any foreseeable risks or discomforts will be discussed with the subject. The protection of confidentiality will be discussed with subjects as well as the subject will be given the name(s)/number(s) of persons to contact should they have any further questions before signing the informed or consent or once they have enrolled in the study. It is reiterated to the subject that participation is voluntary and not participating will not affect present or future medical care. The subject will ask and have answered any and all questions before signing the informed consent. The subject is given a signed copy of the informed consents(s) and HIPAA authorization(s).

MBT testing The ¹³C-Methacetin Breath Test (MBT) is a non-invasive test for assessing liver metabolic function. The BreathID® MCS System consists of the BreathID® MCS device and a test kit containing a breath collection cannula and a non-radioactive isotope 13C-Methacetin solution. It measures and computes the ratio between 13CO2 and 12CO2 in the patient's exhaled breath. The components of the MBT system include the (1MBT BreathID® MCS unit; (2 13C-Methacetin solution. A dedicated flash memory stick for automatic raw data download will be provided to all participating investigative sites. All components of the MBT system will be provided by Exalenz Bioscience Ltd., The MBT BreathID® MCS Unit Exalenz Bioscience Ltd. has developed a molecular correlation spectrometer, based on specific optical-radiation emission and absorption by 13CO2 and 12CO2 gases. This device continuously senses exhaled breath and analyzes CO2 in real-time through a breath collection cannula connected to the patient. Based on Molecular Correlation Spectrometry (MCS), the BreathID® MCS device continuously measures 13CO2 and 12CO2 concentrations from the patient's breath and establishes the 13CO2/ 12CO2 ratio. The cannula continuously transports the breath sample from the patient to the BreathID® MCS device. Depending upon the status of the patient, the cannula may be nasal (for conscious patients) or an adaptor may be used for connection to the ALF-MBT Protocol Page 15 Version 2.0 (19Nov2015) Confidential respiratory line (for intubated patients). Results are displayed in real time on the device screen and are printed after the completion of the test. The BreathID® MCS device calculates the delta over baseline (DOB), which can be translated into the percent dose recovery (PDR) and the cumulative percent dose recovery (CPDR) for each time point derived from the ratio difference compared to baseline (normalized/adjusted to the patient's body weight and height as well as substrate dose) throughout the course of the test. The maximum value of the PDR is called the PDRPeak. The 13C-Methacetin metabolism begins almost immediately since liquid passes through the stomach to the duodenum, where it is absorbed, without delay. The default breath collection test time is one hour after ingestion of 13C-Methacetin. The light sources are 13CO2 and 12CO2 discharging lamps. By using 13CO2 and 12CO2 discharging lamps as light sources, light absorption will be solely due to the existence of 13CO2 and 12CO2 in the gas mixtures. Furthermore, by using 13CO2 and 12CO2 discharging lamps as light sources, background radiation will be substantially reduced, leading to highly sensitive absorption curves. These highly sensitive absorption curves enable detection of very small variations in 13CO2 and 12CO2 concentrations and the 13CO2/ 12CO2 ratio. The BreathID® MCS System can detect variations of less than 1/1000 in the 13CO2/ 12CO2 ratio measurement. The actual breath collection is automatically done by the device and is not operator dependent. If the patient is not connected properly (e.g. the breath does not reach the device), the BreathID® MCS device will prompt the operator to adjust the nasal cannula. The cannula transports the breath sample from the patient to the BreathID® MCS device. The cannula test kit is a single-use kit and is comprised of a plastic sampling line with an in-line hydrophobic filter (used to reduce the amount of moisture present from the patient's breath) and a Luer-lock connector for connection to the BreathID® MCS device. The device is designed to accommodate an extended range of respiratory rates. 3.3.3 13C-Methacetin Exalenz Bioscience Ltd. will supply a ready to use, non-radioactive isotope ¹³C-Methacetin solution for single-use oral administration (75 mg in 150 ml purified water), dispensed in thermoplastic polyester (PTE) bottles sealed with a plastic child resistant stopper. The ¹³CMethacetin solution can be administered via typical oral. 13C-Methacetin meets all of the qualifications for a liver function test substrate: it is a nontoxic small molecule; is administered orally; is rapidly absorbed; and is exclusively metabolized by the liver. Furthermore, 13C can be easily synthesized into a key location within this molecule. No related adverse events have been reported when using this substance, including in vulnerable populations, and the compound remains stable over time. The 13C-Methacetin substrate is a well-known diagnostic reagent that has been described in the literature and used for over 30 years by researchers around the world. ¹³C-Methacetin is rapidly absorbed and metabolized by the hepatic mixed function oxidase, via O-demethylation. This process is carried out by hepatic cytochrome P450 enzymes that produce two products, acetaminophen and formaldehyde, which is transformed through two successive oxidative steps to 13CO2. Toxicology testing results in animals and other clinical information support the safe use of Methacetin in humans. Based on the acute toxicity studies in mice and rats where relatively high LD50 values of 1190mg/kg were administered, the Methacetin dose administered in human breath tests in adults of 75 mg, or approximately 1mg/kg, has a safety ratio in excess of 1000- fold (10). There have been no reports of any complications with the use of this substance in over 2500 patients tested worldwide (see IDE filing). The main metabolite of Methacetin is acetaminophen which has wide routine clinical use at much higher doses than orally administered dose of 13C-Methacetin of 75mg used in this study

Risk Based Monitoring: To ensure compliance with GCP, local regulations and scientific integrity, monitoring of this trial will be managed and oversight retained by the Sponsor or designee.

Requirements for Administration of Substrate: Fasting Subjects will perform the breath test once enrolled into the trial and when the following criteria have been met:

* Oral administration of substrate: The subject should be fasting from solid food for a minimum 6 hours and from oral medications for a minimum of 1 hour
* Subject has not ingested acetaminophen-related medications (e.g. Tylenol) within the past 24 hours (subjects with acetaminophen intoxication may be included 24 hours after ingestion).
* Subject has not had any products containing caffeine for 24 hours.
* Subject has not received general anesthesia in the last 24 hours. Performance of the Breath Collection will be performed after the substrate is administered to the subject; no waiting period is required once the substrate has been administered. Breath is collected automatically via a nasal cannula for a total of 75 minutes (up to 15 minutes for baseline measurement and 60 minutes following ingestion of Methacetin). All test-specific equipment will be supplied by Exalenz

Study Feasibility: The Clinical Research Unit will provide essential resources for the conduct of the proposed research. Study coordinator already experienced form other studies with the Breath ID machine and protocol will be required for administration of the test. Subjects are expected to spend approximately 2 hours in the CRU for administration of MBT test.

Study Limitations: One major limitation to this study is the unknown ability to correlate MBT with various clinical data, specifically variables derived from cardiac catheterization, if not available. Cardiac output, which is measured by cardiac catheterization, is a determinant of hepatic blood flow and likewise, Fontan pressure can influence hepatic perfusion. Cardiac catheterizations are not routinely performed in healthy Fontan patients and any analysis using this variable represents a selection bias towards a symptomatic and potentially sicker subgroup. There is merit in adding a non-invasive test like MBT when looking at FALD patients, given the difficulty to predict liver outcome in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained prior to any study-specific assessments
* Adults patients ≥ 18 years of age
* Liver disease secondary to congenital heart disease or cardiomyopathy

Exclusion Criteria:

* Inability to comprehend and/or give informed consent
* Male and female subjects < 18 years of age
* Females of child-bearing potential that are pregnant or breastfeeding
* Other exclusion criteria include those individuals who are prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-04-21 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2021-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel R Ganger, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] D'Amico G, Garcia-Tsao G, Pagliaro L. Natural history and prognostic indicators of survival in cirrhosis: a systematic review of 118 studies. J Hepatol. 2006 Jan;44(1):217-31. doi: 10.1016/j.jhep.2005.10.013. Epub 2005 Nov 9. No abstract available. PMID 16298014

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the PI's liver/congenital heart disease clinic. Subjects were given details of the study and an IRB approved ICF to review at home. Those interested were later brought in for study visit. They came to the liver clinic for study procedures.
Groups:
- MBT in Liver Disease: Methacetin Breath test (MBT) intervention
  Methacetin Breath Test (MBT): The hypothesis is that MBT CPDR 20 in the Fontan patient is abnormal as a result of alterations in liver perfusion, liver cell metabolic capability and transhepatic resistance secondary to hemodynamics unique to the Fontan as well as end-organ liver damage. Due to lack of robust biomarkers or other risk stratification schemes, we aim to determine whether there is prognostic value in hepatic MBT CPDR 20 in the Fontan patient.
Period: Overall Study
Arm/Group | MBT in Liver Disease
Started | 4 (Four subjects had their first MBT test but due to Covid 19 restrictions unable to return to site for second test.)
Completed | 0 (We did not complete enrollment of 20 subjects as per protocol due to COVID 19 restrictions at our site. Due to covid 19 non-essential procedures were not permitted, in this case the MBT procedure. This limited enrollment and thus we had to close study as we were unable to enroll in a timely manner.)
Not Completed | 4
Not completed — Covid 19 | 4

BASELINE CHARACTERISTICS:
Population: However, with the 4 subjects that we did get baseline data on we have listed results for Breath test (added baseline measure), age, sex, race and region of enrollment.
Groups:
- MBT in Liver Disease: Methacetin Breath test (MBT) intervention
  Methacetin Breath Test (MBT): The hypothesis is that MBT CPDR 20 in the Fontan patient is abnormal as a result of alterations in liver perfusion, liver cell metabolic capability and transhepatic resistance secondary to hemodynamics unique to the Fontan as well as end-organ liver damage. Due to lack of robust biomarkers or other risk stratification schemes, we aim to determine whether there is prognostic value in hepatic MBT CPDR 20 in the Fontan patient.
  Results incomplete as we closed the study due to COVID 19 impacting study recruitment at our site.
Arm/Group | MBT in Liver Disease
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants] — Baseline analysis of age is only based on 4 subjects vs number in protocol as we ended study early due to COVID 19 restrictions. Population: Analysis not performed as study ended early due to Covid 19 pandemic.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 4
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Analysis not performed as study ended early due to Covid 19 pandemic.
  Participants
    Female | 3
    Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Analysis not performed as study ended early due to Covid 19 pandemic.
  Participants
    American Indian or Alaska Native | 0
    Asian | 1
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 3
    More than one race | 0
    Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants] — Population: Analysis not performed as study ended early due to Covid 19 pandemic.
  participants
    United States | 4
Age of participants [Mean (Standard Deviation); unit: years] — Population: Analysis not performed as study ended early due to Covid 19 pandemic.
  years | 36 (9)
PDR (%/hr.) [Mean (Standard Deviation); unit: %/hr.] — Rate at which 13C-Methacetin solution is metabolized, derived from the breath 13C/12C ratio in %/hour
  %/hr. | 35.5 (16.7)
time from administration of 13C methacetin to peak elimination of 13CO2 in mins. [Mean (Standard Deviation); unit: minutes] | 23.7 (12.8)

OUTCOME MEASURES:

1. Primary Outcome: Methacetin Breath Test Results in Patients Undergoing Heart and Liver Transplant Evaluation.
Description: 1. To perform methacetin breath tests (MBT) in a cohort of patients with Congestive (Dilated) Cardiomyopathy and a group of Fontan patients and compare results of the methacetin breath tests to published normal controls. The ¹³C-Methacetin Breath Test (MBT) is a non-invasive test for assessing liver metabolic function. The BreathID® MCS System consists of the BreathID® MCS device and a test kit containing a breath collection cannula and a non-radioactive isotope 13C-Methacetin solution. It measures and computes the ratio between 13CO2 and 12CO2 in the patient's exhaled breath. The components of the MBT system include the 1. MBT BreathID® MCS unit; 2. 13C-Methacetin solution.
  The Cumulative Percent Dose Recovery to be used will be at 20 min (CPDR20) as it correlated with the degree of liver disease severity.
Time Frame: 90 minutes MBT measurement is taken
Population: Per the protocol, 2 MBT tests are required. Due to covid 19 restrictions, subjects could not return for the 2nd test and therefore data analysis could not be performed.
Arm/Group | MBT in Liver Disease
Number analyzed (Participants) | 0

2. Primary Outcome: MR Elastography Results Compared to Methacetin Breath Test Results in Patients Undergoing Heart and Liver Transplant Evaluation.
Description: To explore any association between MBT parameter and clinical parameters available.
  Liver stiffness (using ARFI or MR elastography).
Time Frame: 1 hour for MR elastography
Population: Per protocol, subjects were required to have 2 MBT tests. Due to covid 19 restrictions, subjects could not return to have second required MBT test nor have elastography performed as non-essential procedures were not allowed. This limited enrollment and analysis and therefore, we had to close the study.
Arm/Group | MBT in Liver Disease
Number analyzed (Participants) | 0

3. Primary Outcome: To Explore Any Association Between MBT Parameter and Clinical Parameters Already Available Per Standard of Care in Patients Undergoing Heart and Liver Transplant Evaluation.
Description: To explore any association between MBT parameter and clinical Standard of Care parameters, including Fontan hemodynamics as assessed by either of the following tests: cardiac catheterization, echocardiography, non-invasive imaging of the liver (CT or MRI), non-invasive assessment of liver stiffness (ARFI, MRE or Fibroscan), laboratory investigations, and clinical characteristics (i.e. age of patient, time since Fontan operation, type of Fontan etc., onset of DCM) within 12 months of the study.
  The ¹³C-Methacetin Breath Test (MBT) is a non-invasive test for assessing liver metabolic function. The BreathID® MCS System consists of the BreathID® MCS device and a test kit containing a breath collection cannula and a non-radioactive isotope 13C-Methacetin solution. It measures and computes the ratio between 13CO2 and 12CO2 in the patient's exhaled breath. The components of the MBT system include the 1. MBT BreathID® MCS unit; 2. 13C-Methacetin solution.
Time Frame: 1 year
Population: Due to covid 19 restrictions subjects did not complete procedures so could not analyze data as per protocol. Note I have to add primary measure above otherwise I get errors. The primary measure could not be analyzed so I am putting 0 in the arms/group and outcome measure table since no analysis.
Arm/Group | MBT in Liver Disease
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were monitored, but none observed, for 1 year for subject total participation. Per protocol, subjects would have been observed for 3-5 years during the study. However due to COVID 19 restrictions at our site study was unable to complete a second MBT test on subjects that were enrolled. So we were unable to complete the study as no subjects returned for a second test.
Description: Adverse events were monitored for the first year of the study in the 4 enrolled subjects, but none observed.
Groups:
- MBT in Liver Disease: Methacetin Breath test (MBT) intervention on patients undergoing heart and liver transplant evaluation
Arm/Group | MBT in Liver Disease
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
Due to COVID 19 restrictions at our site study could not be completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-11-15): https://cdn.clinicaltrials.gov/large-docs/58/NCT04176458/Prot_002.pdf